CLINICAL TRIAL: NCT03981393
Title: Cardinality Matching Study of Early v.s. Delayed VV ECMO in Severe Respiratory Failure
Status: Completed | Type: Observational
Sponsor: University of Cambridge (Other)
Responsible Party: Principal Investigator, Alex Warren, Academic Foundation Doctor, University of Cambridge
Other Study IDs: ECMO-002
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Respiratory Failure; ECMO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 'Less severe hypoxaemia': PaO2/FiO2 ratio > 68 mmHg (9.1kPa) at decision-to-cannulate
- 'Very severe hypoxaemia': PaO2/FiO2 ratio ≤ 68 mmHg (9.1kPa) at decision-to-cannulate

SUMMARY:
Clinical reasoning and recent data suggest that early use of venovenous extracorporeal membrane oxygenation in refractory respiratory failure may confer a survival advantage.

This retrospective matched study will assess whether patients who received VV ECMO at less severe hypoxaemia had differing outcomes to those who received ECMO with very severe hypoxaemia.

DETAILED DESCRIPTION:
VV ECMO is increasingly used in refractory respiratory failure. Despite advances in lung protective ventilation strategies, patients who have severe respiratory failure often develop complications from mechanical ventilation, including volutrauma and barotrauma. ECMO allows gas exchange to occur extracorporeally and may reduce the potential burden of iatrogenic lung injury by allowing a reduction of volume and pressure support - a 'lung rest' strategy. It is theorised that earlier intitiation of ECMO may allow for better outcomes, as there will have been less time for iatrogenic lung injury to occur.

The UK ECMO registry has been collected of patients treated under the NHS England commissioned respiratory ECMO service since 2011. This study has been previously registered and publication is intended shortly.

Patients will be extracted from this registry if they received VV ECMO. Propensity matching scores will be created and patients will be stratified into groups of 'early' vs 'delayed' ECMO, based on their probability of being in either group.

Patients will be divided into cohorts based on the median PaO2/FiO2 ratio at decision to cannulate ('less severe hypoxaemia') and ('very severe hypoxaemia'). Matched cohorts will be created correcting for key confounding factors (age, primary diagnosis, duration of pre-ECMO ventilation and PaCO2), using cardinality matching (a novel technique described by Zubizaretta et al. in 2014) and traditional propensity-score-based methods.

The technique with greater balance and statistical power (as defined by sample size) will be selected for the primary analysis.

Further analyses will assess the relationship between hypoxaemia at decision-to-cannulate and confounding factors as above.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the UK ECMO registry (see previous registration; NCT number awaited; protocol ECMO-001)
* Patients with VV ECMO

Exclusion Criteria:

* Patients with inadequate or missing data for creation of propensity score models.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prespecified secondary analysis of the UK ECMO registry. Inclusion criteria are ultimately at the discretion of each recruiting centre, but includes adult patients with potentially reversible acute respiratory failure without absolute contraindications to ECMO therapy.
Sampling Method: Non-Probability Sample
Enrollment: 667 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Survival to ECMO ICU discharge | Up to 90 days.
  Percentage of patients alive at discharge from the ICU at the specialist ECMO centre

SECONDARY OUTCOMES:
Duration of ECMO treatment | Up to 90 days.
  Duration spent supported by active ECMO treatment.

IPD SHARING:
Plan to Share IPD: Undecided
Access to IPD is via the UK ECMO network steering group. Enquiries in the first instance can be made to Dr Alain Vuylsteke, at a.vuylsteke@nhs.net